CLINICAL TRIAL: NCT01835743
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia HP Scanner (HPS) Laser on Chronic Heel Pain
Brief Title: Study of Low Level Laser Therapy to Treat Chronic Heel Pain Arising From Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_HP_001
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia HPS Laser (Active Comparator): The Erchonia HPS Laser contains 3 independent diodes mounted in scanner devices and positioned equidistant from each other and titled at a 30 degree angle. Each scanner emits 17 milliwatts (mW), 635 nm of red laser light.
  Interventions: Device: Erchonia HPS Laser
- Placebo Laser (Placebo Comparator): The Placebo Laser is identical in appearance and operation to the Erchonia HPS Laser but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia HPS Laser — The Erchonia HPS Laser is administered to the subject's heel 6 times across 3 consecutive weeks, 2 times each week, for 10 minutes of treatment time per administration.
  Arms: Erchonia HPS Laser
Device: Placebo Laser — The Placebo Laser is administered to the subject's heel 6 times across 3 consecutive weeks, 2 times each week, for 10 minutes of treatment time per administration.
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether the Erchonia HPS Laser is effective in the treatment of chronic heel pain arising from plantar fasciitis.

DETAILED DESCRIPTION:
Chronic heel pain is one of the most common forms of foot pain in adults. The heel bone (calcaneus) receives a lot of stress as it is the largest bone in the foot, and the heel is the first part of the foot to contact the ground during walking. Normally, as the foot absorbs the weight of the body during walking, the arch area joint locking mechanism provides about 80% of the stability of the foot. The other 20% of biomechanical stability is provided by the plantar fascia and muscles, tendons, and ligaments. Gait abnormalities can cause inflammation of the structures attached to the heel bone, resulting in heel pain.

Plantar fasciitis refers to syndromes of pain that occurs at the site of the attachment of the plantar fascia and the calcaneus, with or without accompanying pain along the medial band of the plantar fascia. Eighty per cent (80%) of heel pain is caused by plantar fasciitis, with 10% of the U.S. population likely to be afflicted over a lifetime. Two million Americans are treated for plantar fasciitis each year. It is more common in women than men and in people aged 40-60 years.

Plantar fasciitis results from small tears and inflammation in the wide band of tendons and ligaments that stretch from the heel to the ball of the foot. This band forms the arch of the foot and serves as a shock absorber for the body. Causes of plantar fasciitis include poor footwear, sedentary lifestyles, obesity and sports injuries. Plantar fasciitis is characterized by pain at the bottom of the heel on weight bearing, particularly when first arising in the morning, and after prolonged periods of rest.

Progressive conservative treatment options for plantar fasciitis include rest, stretching, strengthening, massage, physical therapy, orthotics and shoe inserts, heel cups, night splints, plantar strapping, non-steroidal anti-inflammatories (NSAIDs), steroid and corticosteroid injections and iontophoresis. When conservative treatments are unsuccessful, surgical release or removal of the plantar fascia may occur.

However, most conservative approaches are of limited effectiveness and there are potential significant complications from plantar fascia surgery.

Low level laser therapy (LLLT) offers a quick, painless, non-invasive, side-effect free alternative to relieve the debilitating pain of plantar fasciitis. When applied to injuries and lesions, low level laser light has been shown to stimulate healing and reduce pain by accelerating the speed, quality and strength of tissue repair and the reduction of inflammation. Laser therapy has been found to be particularly effective over other standard therapies in relieving pain and other symptoms associated with chronic problems and injuries as it impacts the complete system of targeted muscles, tendons, ligaments, connective tissue, bone, nerve, and dermal tissues. Additionally, Erchonia low level lasers have been shown through controlled clinical trials to be effective for pain reduction, as evidenced through several FDA 510(k) approvals for various indications.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral mechanical plantar heel pain
* Chronic heel pain defined as at least 3 months of ongoing heel pain with no evidence of acute trauma to the heel
* Degree of heel pain rating on the 0-100 Visual Analog Scale (VAS) is at least 50 for heel pain experienced upon taking the first few steps of the day.
* Heel pain has been previously unresponsive to prescription non-steroidal anti-inflammatory drugs (NSAIDs) taken over a minimum period of 2 weeks; and any two or more of the following conservative treatments: rest, taping, stretching, orthotics, shoe modifications, night splinting, casting, physical therapy, or local corticosteroid injections
* Subject is willing and able to refrain from consuming non-study approved medications or partaking in other therapies for relief of heel pain throughout study participation

Exclusion Criteria:

* Inability to definitively rule out any one or more of the following potential etiologies of chronic heel pain: mechanical posterior; neurologic; arthritic; and traumatic heel pain
* Bilateral heel pain
* Evidence of acute trauma to the heel
* Loss of plantar foot sensation
* Foot deformity
* Previous surgery to the heel
* Foot trauma within the previous three months
* Skin ulceration (infection or wound) on the heel and surrounding area
* Sciatica
* Benign and malignant tumors
* Acute infection of soft tissue or bone such as osteomyelitis
* Diabetic neuropathic pain
* Type I Diabetes
* Sensory neuropathy
* Previous diagnosis of neuropathy affecting lower extremities
* Peripheral vascular disease or autoimmune disease
* Fibromyalgia
* Chronic fatigue syndrome
* Chronic pain disorders
* Metabolic disorders: Osteomalacia, Paget's disease, Sickle cell disease.
* Blood coagulation disorders
* Significant heart conditions including coronary heart failure (CHF) and implantable heart devices
* Non-ambulatory status
* Unable or unwilling to consume the study rescue medication of Tylenol
* Photosensitivity disorder
* Pregnant or lactating
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the consent form or the ability to record the study measures
* Involvement in litigation or a worker's compensation claim or receiving disability benefits related to the heel pain
* Participation in other research in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Coughlin, M.D., Principal Investigator; Kerry Zang, D.P.M., Principal Investigator
Locations (2):
- United States (2):
  - Arizona Institute of Footcare Physicians, Mesa, Arizona
  - Coughlin Foot and Ankle Clinic, Boise, Idaho

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia HPS Laser | Placebo Laser
Started | 37 | 32
Completed | 37 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia HPS Laser | Placebo Laser | Total
Number analyzed (Participants) | 37 | 32 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.70 (10.46) | 55.81 (12.33) | 56.29 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 34 | 29 | 63
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 32 | 69
Heel Side [Number; unit: participants] — Heel side (right heel or left heel) that qualified for and received the study procedure administrations
  participants
    Right Heel | 20 | 9 | 29
    Left Heel | 17 | 23 | 40
Duration of Heel Pain at Baseline [Mean (Standard Deviation); unit: months] — The duration of heel pain at baseline was recorded as subject reported length of experiencing heel pain to that timepoint, in months.
  months | 12.34 (11.08) | 12.23 (12.41) | 12.29 (11.63)
Degree of Heel Pain at Baseline [Mean (Standard Deviation); unit: units on a scale] — Subjects rated the overall degree of pain experienced in the heel region of the heel being treated and evaluated in the study upon waking in the morning and taking the first few steps of the day for 2 consecutive days before receiving the first study procedure with the Erchonia HPS. The degree of pain was recorded by placing a cross along the point that best represented their current heel pain level on the 0-100 mm (0 -10 cm) Visual Analog Pain Scale (VAS) ranging from '0: no pain at all' to '100: worst pain imaginable,'. The higher the rating, the greater the heel pain experienced.
  units on a scale | 69.15 (12.65) | 67.70 (11.80) | 68.48 (12.19)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Attained a Change of -30% or Greater in the VAS Score
Description: Each subject rated heel pain upon taking the first few steps of the day on the 0-100 mm (0 -10 cm) Visual Analog Pain Scale (VAS) from '0: no pain at all' to '100: worst pain imaginable'. The higher the VAS score, the greater the heel pain experienced. Percent (%) change in VAS score was calculated as the % difference in VAS score at week 5 (2 weeks after procedure administration end) relative to baseline evaluation. A negative (-) % difference in VAS score across the evaluation period indicated a decrease (improvement) in heel pain, and a positive (+) % difference in VAS score indicated an increase (worsening) in heel pain. A change of -30% or greater in the VAS score was considered positive for study success. The number of participants who attained a change of -30% of greater in VAS score across the evaluation period was calculated for both subjects in the test group and in th placebo group as a proportion of the total number of subjects in each procedure group.
Time Frame: baseline and 5 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia HPS Laser | Placebo Laser
Number analyzed (Participants) | 37 | 32
participants | 23 | 4
Statistical Analysis 1: Comparison: Erchonia HPS Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.00005, Fisher Exact

2. Secondary Outcome: Change in Heel Pain Score on the Visual Analog Scale (VAS)
Description: Each subject rated heel pain upon taking the first few steps of the day on the 0-100 mm (0 -10 cm) Visual Analog Pain Scale (VAS) from '0: no pain at all' to '100: worst pain imaginable'. The higher the VAS score, the greater the heel pain experienced. Change in heel pain score on the VAS was calculated as the heel pain VAS score at week 5 (2 weeks after procedure administration end) minus the heel pain VAS score at baseline evaluation. A negative (-) change in heel pain VAS score across the evaluation period indicated a decrease (improvement) in heel pain and was positive for study success. A positive (+) change in heel pain VAS score indicated an increase (worsening) in heel pain and was negative for study success.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: scores on a 0-100 VAS scale
Arm/Group | Erchonia HPS Laser | Placebo Laser
Number analyzed (Participants) | 37 | 32
scores on a 0-100 VAS scale | -29.47 (24.94) | -5.38 (16.01)
Statistical Analysis 1: Comparison: Erchonia HPS Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; t-test for two independent samples to compare the change in VAS scores across the evaluation period between the two procedure administration groups

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Erchonia HPS Laser | Placebo Laser
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 0/37 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No